CLINICAL TRIAL: NCT06760962
Title: Reflective Mindfulness and Emotional Regulation Training to Enhance Nursing Students' Self-Awareness, Understanding, and Regulation: a Mixed Method Randomized Controlled Trial
Brief Title: Reflective Mindfulness and Emotional Regulation Training to Enhance Nursing Students' Self-Awareness, Understanding, and Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed El-Ashry, Lecturer, PhD, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Nursing college, Benha Univ
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Undergraduate Health Professional Students
Keywords: Mindfulness; emotional regulation; nursing students; nursing education; self-awareness; mixed method
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The RMERT program consisted of six weekly 90-minute sessions facilitated by researchers trained in cognitive behavioral therapy (CBT) and transactional analysis (TA). The training employed the ABC model of CBT (Activating events, Beliefs, and Consequences) to address maladaptive cognitive patterns, along with TA techniques such as empathic inquiry and reflection. Relaxation strategies, including diaphragmatic breathing and progressive muscle relaxation, were also integrated. The sessions focused on enabling students to reflect on their mental and emotional states, process their feelings, and apply cognitive reappraisal-a healthy emotional regulation strategy-instead of relying on expressive suppression, which is maladaptive.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Forty students met the eligibility requirements and were randomly assigned at a 1:1 ratio to control and intervention groups of twenty each. The intervention set was then split into ten subgroups to form counseling groups. The intervention and control groups completed the pre-test and post-tests one week before the sessions began and one week after they ended. Students' identifiers were removed to ensure confidentiality. In two subgroups of 10, each intervention group attended intervention sessions, while the control group did not receive any intervention sessions. During the intervention sessions, both groups attended the theoretical and clinical parts of the psychiatric mental health nursing course with their colleagues. As part of their training, they facilitated nursing services for actual patients in clinical settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental)
  Interventions: Behavioral: Reflective Mindfulness and Emotional Regulation training
- control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Reflective Mindfulness and Emotional Regulation training — The RMERT program consisted of six weekly 90-minute sessions facilitated by researchers trained in cognitive behavioral therapy (CBT) and transactional analysis (TA). The training employed the ABC model of CBT (Activating events, Beliefs, and Consequences) to address maladaptive cognitive patterns, along with TA techniques such as empathic inquiry and reflection. Relaxation strategies, including diaphragmatic breathing and progressive muscle relaxation, were also integrated. The sessions focused on enabling students to reflect on their mental and emotional states, process their feelings, and apply cognitive reappraisal-a healthy emotional regulation strategy-instead of relying on expressive suppression, which is maladaptive.
  Arms: study group

SUMMARY:
This study assessed the impact of a six-week Reflective Mindfulness and Emotional Regulation Training (RMERT) program on fourth-year nursing students. Using a randomized controlled trial with 40 participants, the intervention group (n=20) received RMERT, while the control group (n=20) continued standard coursework.

DETAILED DESCRIPTION:
This study evaluated the effectiveness of Reflective Mindfulness and Emotional Regulation Training (RMERT) in enhancing nursing students' self-awareness, emotional understanding, and regulation. Nursing students frequently face significant academic and psychological challenges, particularly in mental health nursing courses, which can lead to stress, anxiety, and compromised well-being. RMERT was designed as a psychoeducational intervention integrating mindfulness and emotional regulation techniques to help students develop critical skills for managing these challenges.

Study Design The randomized controlled trial employed a mixed-methods approach and involved 40 fourth-year undergraduate nursing students at Benha University. Participants were randomly allocated into an intervention group (n=20) and a control group (n=20). The intervention group attended a six-week RMERT program, while the control group continued their standard academic activities without additional interventions. Both groups underwent pre- and post-intervention assessments using validated instruments: the Emotion Regulation Questionnaire (ERQ) and the Mindful Attention Awareness Scale (MAAS). Qualitative data, collected exclusively from the intervention group, were analysed thematically.

Intervention The RMERT program consisted of six weekly 90-minute sessions facilitated by researchers trained in cognitive behavioural therapy (CBT) and transactional analysis (TA). The training employed the ABC model of CBT (activating events, beliefs, and consequences) to address maladaptive cognitive patterns, along with TA techniques such as empathic inquiry and reflection. Relaxation strategies, including diaphragmatic breathing and progressive muscle relaxation, were also integrated. The sessions focused on enabling students to reflect on their mental and emotional states, process their feelings, and apply cognitive reappraisal-a healthy emotional regulation strategy-instead of relying on expressive suppression, which is maladaptive.

ELIGIBILITY:
Inclusion Criteria:

* Students enroled in the psychiatric/mental health nursing course for the first time, i.e., did not enrol in or join similar or the same course before.
* for example, joined the faculty from the secondary school, not through other paths or bridging educational programs that would include psychiatric/mental health courses/modules as part of their programs
* did not fail the course before or attended it for more time.

Exclusion Criteria:

no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire | 6 weeks
  Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores in each subscale. The higher the score, the greater the use of that strategy and vice-versa.
The Mindful Attention Awareness Scale (MAAS) | 6 weeks
  The Mindful Attention Awareness Scale (MAAS), developed by Brown and Ryan in 2003, is a 15-item self-report instrument designed to measure a fundamental aspect of mindfulness: a receptive and attentive state of awareness focused on the present moment. Respondents rate their experiences using a six-point Likert scale, ranging from 1 ("almost always") to 6 ("rarely"). The MAAS has demonstrated strong psychometric properties and has been validated across diverse populations, including college students, community members, and individuals with cancer. The overall score is calculated as the average of the 15 items, with higher scores reflecting greater mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of nursing Alexandria university, Alexandria, None Selected, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study authors indicated that individual participant data (IPD), including the following, will be shared upon reasonable request:
  De-identified Data:
  Pre- and post-intervention scores from the Emotion Regulation Questionnaire (ERQ) and the Mindful Attention Awareness Scale (MAAS).
  Demographic and baseline data (e.g., age, gender, residence, GPA, marital status, and employment status) in de-identified format.
  Qualitative Data:
  De-identified transcriptions of intervention group sessions used for thematic analysis.
  Study Protocol and Analysis Plans:
  The detailed intervention framework, including the six-session RMERT program outline.
  Quantitative and qualitative data analysis plans.
  Consent Documentation:
  Sample forms used to obtain participant consent (in anonymized form).
  Ethical Approvals:
  Approval details are provided by the Research Ethics Committee. This data will be made available upon request to the corresponding author, provided the request aligns with ethical considerations.
Supporting Information: Study Protocol
Time Frame: 2 weeks
Access Criteria: all authors of the study

REFERENCES:
- [Background] Veigh CM, Reid J, Carswell C, Ace L, Walsh I, Graham-Wisener L, Rej S, Potes A, Atkinson K, Edginton T, Noble H. Mindfulness as a well-being initiative for future nurses: a survey with undergraduate nursing students. BMC Nurs. 2021 Dec 20;20(1):253. doi: 10.1186/s12912-021-00783-0. PMID 34930234
- [Background] McVeigh C, Ace L, Ski CF, Carswell C, Burton S, Rej S, Noble H. Mindfulness-Based Interventions for Undergraduate Nursing Students in a University Setting: A Narrative Review. Healthcare (Basel). 2021 Nov 2;9(11):1493. doi: 10.3390/healthcare9111493. PMID 34828538
- [Derived] Salem GMM, Hashimi W, El-Ashry AM. Reflective mindfulness and emotional regulation training to enhance nursing students' self-awareness, understanding, and regulation: a mixed method randomized controlled trial. BMC Nurs. 2025 Apr 30;24(1):478. doi: 10.1186/s12912-025-03086-w. PMID 40307764